CLINICAL TRIAL: NCT03880123
Title: A Phase I Study of the Selective Inhibitor of Nuclear Export (SINE) Selinexor in Combination With the Proteasome Inhibitor Ixazomib for the Treatment of Advanced Sarcoma
Brief Title: Selinexor in Combination With Ixazomib for the Treatment of Advanced Sarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study will not proceed, no participants enrolled.
Sponsor: Matthew Ingham (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Matthew Ingham, Assistant Professor of Medicine (Oncology), Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS0199
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Liposarcoma; Malignant Peripheral Nerve Sheath Tumors; Alveolar Soft Part Sarcoma; Ewing Sarcoma; Sarcoma
Keywords: Liposarcoma; Malignant Peripheral Nerve Sheath Tumors; Alveolar Soft Part Sarcoma; Ewing Sarcoma; Selinexor; ixazomib; sarcoma; kpt-330
MeSH Terms: conditions — Liposarcoma; Neurofibrosarcoma; Sarcoma, Alveolar Soft Part; Sarcoma, Ewing; Sarcoma | interventions — selinexor; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor/Ixazomib (Experimental): Patients will receive combination treatment with selinexor and ixazomib. The dose of ixazomib is fixed at 4 mg, whereas several different dose levels of selinexor may be evaluated. No patients will receive a placebo.
  Interventions: Drug: Selinexor; Drug: Ixazomib

INTERVENTIONS:
Drug: Selinexor — Selinexor will be taken orally on Days 1, 8, 15, and 22 of each cycle at the following dose levels (DLs):
  DL 1: 40 mg; DL 2: 60 mg; DL 3: 80 mg; DL 4: 100 mg
  The selinexor product is provided as 20 mg tablets in wallet-sized blister packs. Selinexor should be taken together with ixazomib.
  Other Names: KPT-330
Drug: Ixazomib — Ixazomib will be taken orally on Days 1, 8, and 15 of each cycle at the same dose level: 4 mg.
  The ixazomib product is provided in strengths of 4.0, 3.0, and 2.3 mg capsules as the active boronic acid. Ixazomib should be taken on an empty stomach (no food or drink) at least 1 hour before or at least 2 hours after food.
  Other Names: Ninlaro

SUMMARY:
The main purpose of this study is to establish a safe and tolerable dose combination (the "maximum tolerated dose") of selinexor and ixazomib when used together for the treatment of patients with certain types of advanced sarcoma. The study will enroll patients with advanced dedifferentiated liposarcoma, malignant peripheral nerve sheath tumor, alveolar soft part sarcoma and Ewing sarcoma. Future studies to further evaluate the safety and anti-cancer efficacy of this treatment for sarcoma will use the dose combination determined in this study.

DETAILED DESCRIPTION:
Sarcoma is a rare form of cancer which originates from the soft tissues and bones of the body. There are more than 50 different types of sarcoma. The primary treatment approach for most types of advanced sarcoma involves chemotherapy, but newer treatment approaches are needed because chemotherapy is not curative, sometimes does not work well, and often has significant side effects.

The purpose of this study is to evaluate a new treatment for certain types of sarcoma. The new treatment involves two oral targeted drugs used in combination: selinexor and ixazomib. Selinexor inhibits the transport of certain proteins between the nucleus and the cytoplasm of the cell. Ixazomib is part of a class of drugs called proteasome inhibitors. Currently, neither of these drugs is approved for the treatment of sarcoma. The researchers believe this combination treatment may work effectively for certain types of sarcoma based on encouraging laboratory research results. The types of sarcoma in which the treatment will be tested are: dedifferentiated liposarcoma, alveolar soft part sarcoma, malignant peripheral nerve sheath tumor, and Ewing sarcoma. The purpose of this study is to define doses of selinexor and ixazomib that are safe and tolerable for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age ≥ 14 years
3. Body surface area ≥ 1.2 m2
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Histologically confirmed de-differentiated liposarcoma, malignant peripheral nerve sheath tumor, alveolar soft part sarcoma or Ewing sarcoma. Liposarcomas with areas of well-differentiated disease are eligible if there is a biopsy-proven component of dedifferentiated liposarcoma. Pathology is reviewed at Columbia University Medical Center.
6. Disease which is locally advanced and unresectable or metastatic. Disease which may be resected but with an associated level of morbidity deemed unacceptable by the treating clinician is considered eligible.
7. Measurable disease as assessed by RECIST criteria version 1.1.
8. Progression on, or intolerance to, at least one prior systemic regimen for sarcoma (including systemic treatment used in the adjuvant or neoadjuvant settings). For alveolar soft part sarcoma and dedifferentiated liposarcoma, there is no upper limit on the number of prior therapies that may have been received. For Ewing sarcoma and malignant peripheral nerve sheath tumor, patients may have received no more than 3 prior lines of therapy (excluding systemic treatment used in the adjuvant or neoadjuvant settings).
9. Acceptable organ and marrow function as defined below:

   Absolute neutrophil count (ANC) ≥ 1,500/mm3 Hemoglobin ≥ 8.5 g/dL Platelet count ≥ 100,000/mm3 Calculated creatinine clearance > 30 mL/min Total bilirubin ≤ 1.5 times upper limit of normal Aspartate Transaminase (AST) /Alanine Transaminase (ALT) ≤ 3.0 times upper limit of normal
   * Upper limit of normal is defined by the clinical laboratory performing the test.
   * Creatinine clearance is obtained using the lean body mass formula (Modified Cockcroft Gault)
   * If transaminase elevation and/or bilirubin elevation is attributed to the presence of liver metastases, a total bilirubin ≤ 2.5 times the upper limit of normal and an Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤ 2.5 times the upper limit of normal are permissible. Patients with an elevated bilirubin level that is attributed to an inherited disorder, such as Gilbert's disease, may be enrolled at the discretion of the principal investigator.
   * Patients may not receive platelet transfusions within 3 weeks of initiating protocol therapy.
10. Meet the following criteria regarding contraception:

Female patients who:

1. Are postmenopausal for at least 1 year before the screening visit, OR
2. Are surgically sterile, OR
3. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
4. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Male patients who: (must meet criteria even if surgically sterilized, i.e. after vasectomy):

1. Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

1. Received selinexor or another XPO1 inhibitor previously.
2. Received ixazomib or another proteasome inhibitor previously.
3. Currently pregnant or lactating.
4. Prior malignancy that required treatment, or has shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) during the 5 years prior to registration. Cancer treated with curative intent more than 5 years previously and without evidence of recurrence is not an exclusion.
5. Received any systemic anticancer therapy including investigational agents or radiation ≤3 weeks (or ≤5 half-lives of the drug, whichever is longer) prior to registration. Patients must have recovered to grade ≤ 1 or baseline from clinically significant adverse effects associated with prior anti-cancer therapies except for alopecia or controlled endocrinopathies.
6. Major surgery within 2 weeks of first dose of study treatment.
7. Any serious medical or psychiatric illness, medical condition or organ dysfunction which, in the investigator's opinion, could compromise patient safety or compliance with the protocol.
8. Unstable cardiovascular function as defined by:

   1. Symptomatic ischemia, or
   2. Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmia are excluded; 1st degree arterioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
   3. Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥3, or
   4. Myocardial infarction (MI) within 6 months
9. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment. Prophylactic use of antibiotics and/or antivirals is acceptable.
10. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positivity.
11. History of clinically significant ocular disease manifest by visual defects or disturbances, including those caused by active glaucoma or cataracts, which have not been addressed by surgery or other corrective intervention. If necessary, an opthalmologic exam should be performed at screening.
12. Inability to swallow tablets, clinically significant malabsorption syndrome, or any other GI disease or dysfunction that could interfere with absorption of study drugs.
13. Presence of grade 3 peripheral neuropathy or grade 2 peripheral neuropathy with pain at any time during the screening period.
14. Systemic treatment, within 14 days before initiation of study treatment, with strong CYP3A4 inducers (including, but not limited to rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or use of St. John's wort.
15. Unwillingness to comply with the study protocol and/or procedures.
16. Central nervous system involvement.
17. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
18. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 2 years
  To establish the maximum tolerated dose combination for selinexor and ixazomib when used as a combination treatment for patients with dedifferentiated liposarcoma, malignant peripheral nerve sheath tumor, alveolar soft part sarcoma and Ewing sarcoma. The MTD is defined by the time to event continual reassessment method, a model-based dose finding study design.

SECONDARY OUTCOMES:
Adverse Event (AE) Rate | Up to 2 years
  Adverse events will be collected from the day the patient receives the first dose of study treatment until 30 days after end-of-treatment. Adverse events will be reported by Common Terminology Criteria for Adverse Events (CTCAE criteria), stratified by grade.

OTHER OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  The percentage of patients who experience a partial or complete response to study therapy as assessed radiographically by RECIST version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ingham, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No